CLINICAL TRIAL: NCT04359381
Title: Kinesiotaping Versus Pilate Exercises on Primary Dysmenorrhea
Brief Title: Kinesiotaping Versus Pilate Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Amira Hassan Abdelaziz (Unknown); Soheir Mahmoud El-Kosery (Unknown)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, assistant professor Department of Physical Therapy for Women's Health, Faculty of Physical therapy, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Dysmenorrhea; Exercise
Keywords: kinesiotaping; pilate exercises; primary dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomized controlled trial.
Who Masked: Investigator
Masking Description: An independent person randomly assigned to all participated subjects to either group (A) (n=30) or group (B) (n=30) by chosen numbers from closed envelopes having numbers that the number generator were chosen randomly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotaping (Experimental): by kinesiotaping during menstruation for 3 successive menstruation
  Interventions: Other: kinesiotaping application
- pilate exercises (Experimental): pilate exercises, 3 sessions per week for 3 months
  Interventions: Other: Pilate exercises program

INTERVENTIONS:
Other: kinesiotaping application — kinesiotaping was applied once the menstrual pain begins (one day before menstruation) for periods of 4 to 5 days until the pain disappears and then removed it. Kinesiotaping was used for 3 successive menstruations.
  Arms: kinesiotaping
Other: Pilate exercises program — Each girl in group (B) was engaged in a supervised pilate exercises program for 30 minutes per session for 3 days/week for 12 weeks except days of menstruation. Participants would be oriented to wear comfortable clothes .
  Arms: pilate exercises

SUMMARY:
Sixty girls participated in this study and their main complaints were pain and cramping during menstruation. They were divided randomly into two equal groups.

DETAILED DESCRIPTION:
Group (A) (30 girls) treated by kinesiotaping during menstruation for 3 successive menstruation. Group (B) (30 girls) treated by pilate exercises, 3 sessions per week for 3 months except the days of menstruation. Visual analogue scale to assess pain intensity, Quality of life enjoyment and satisfaction questionnaire, Menstrual Distress Questionnaire, WALIDD score, Spielberger questionnaire and blood sample analysis to estimate plasma prostaglandin level were applied for each girl in both groups before and after the treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Their ages ranged from 14 to 20 years old
* their body mass index (BMI) would be less than 25 Kg/m2
* having primary dysmenorrhoea

Exclusion Criteria:

* skin diseases or cardiac diseases
* irregular or infrequent menstrual cycles
* previous abdominal or back operations

Ages: 14 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Weight and height scale | three months
  Was used to measure the weight and height of each girl before starting the study and to calculate BMI according to the following formula: BMI = weight (kg) / height square (m)2

SECONDARY OUTCOMES:
Visual analog scale | three months
  For determining pain intensity before and after the treatment course for each girl in both groups (A&B). VAS is a-10 cms line, at one end was written (no pain = zero) and at the other end was written (worst pain the patient ever felt = 10)

CONTACTS AND LOCATIONS:
Overall Officials: ghada eb elrefaye, professor, Principal Investigator — Assistant Professor of Physical Therapy for Woman's Health, Cairo University
Locations (1):
- Ghada Elrefaye, Cairo, Egypt